CLINICAL TRIAL: NCT02794714
Title: Comparing Deep Neuromuscular Block and Moderate Neuromuscular Block in Patients Undergoing Laparoscopic Gynaecological Surgeries: Impact on Surgical Satisfaction of Operating Conditions and Patient Satisfaction
Brief Title: Deep vs Moderate Block: Impact on Operating Conditions & Patient Satisfaction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: unresolved budget issues
Sponsor: Kuala Lumpur General Hospital (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Loo Su Yin, Dr, Kuala Lumpur General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVL#123
Record Dates: First submitted 2016-05-19; First posted 2016-06-09 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Neuromuscular Blockade
Keywords: Laparoscopic Gynecologic Surgeries
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- deep neuromuscular blockade (Experimental): Rocuronium will be administered to achieve PTC 1-2 throughout surgery.
  Interventions: Drug: Moderate neuromuscular blockade
- moderate neuromuscular blockade (Active Comparator): Rocuronium will be administered to achieve TOFC 2 throughout surgery
  Interventions: Drug: Deep neuromuscular blockade

INTERVENTIONS:
Drug: Deep neuromuscular blockade — Deep neuromuscular blockade attained during surgery using Rocuronium 0.6mg/kg at induction of anesthesia with intermittent boluses of 0.15 - 0.2 mg/kg to maintain a Post Tetanic Count (PTC) of 1-2 throughout surgery. Neuromuscular blockade reversed at the end of surgery with Sugammadex 4mg/kg.
  Other Names: Rocuronium, Esmeron
  Arms: moderate neuromuscular blockade
Drug: Moderate neuromuscular blockade — Moderate neuromuscular blockade attained during surgery using Rocuronium 0.6mg/kg at induction with intermittent boluses of 0.15 - 0.2 mg/kg to maintain Train of Four Count (TOFC) of 2 throughout surgery. Neuromuscular blockade reversed at the end of surgery with Sugammadex 2mg/kg.
  Other Names: Rocuronium, Esmeron
  Arms: deep neuromuscular blockade

SUMMARY:
This study compares surgeon's satisfaction of operating conditions and patient's satisfaction following laparoscopic gynecological surgeries in two groups of patients, half of whom will receive deep neuromuscular blockade and the other half, moderate neuromuscular blockade.

DETAILED DESCRIPTION:
Deep neuromuscular blockade in anesthesia has been shown to improve operating conditions in retroperitoneal surgeries, while there is minimal evidence regarding this method in laparoscopic gynecological procedures.The advantage of improving surgical conditions with a deep neuromuscular blockade in laparoscopic surgery may however lead to a delayed neuromuscular recovery and hence a delay in turnover of patients.

Rocuronium will be used for muscle relaxation in order to achieve the necessary depth of neuromuscular blockade. Sugammadex is a modified cyclodextrin that forms complexes with rocuronium, reducing free plasma concentrations of rocuronium and reversing its neuromuscular blocking action from any depth.

The use of rocuronium will therefore aid in achieving a deep neuromuscular blockade which the investigators postulate will improve surgical conditions and the reversal with sugammadex will ensure a rapid recovery thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients identified from the anaesthetic clinic scheduled to undergo a laparoscopic gynaecological procedure under general anaesthesia

   * requiring tracheal intubation
   * elective surgeries (eg. laparoscopy & dye insufflation, bilateral tubal ligation, cystectomy, myomectomy, hysterectomy, salpingo-oophorectomy)
2. American Society of Anaesthesiology (ASA) I-II

Exclusion Criteria:

1. Anticipated difficult airway
2. Patients requiring rapid sequence induction
3. Patient anticipated to require admission to the intensive care unit (ICU) or not planned for extubation
4. Patient with liver or renal failure (creatinine clearance <50mls/min)
5. Patients with a baseline heart rate <50/min
6. Patients with documented or suspected neuromuscular disorder

   * Guillain - Barre syndrome
   * Cerebrovascular accidents with residual neurology
   * Parkinson's Disease
   * Myasthenia Gravis
7. Any condition making the administration of patient satisfaction questionnaire difficult/impossible

   • speech or hearing impairment and language barriers
8. Patients on fusidic acid or toremifene 24 hours before surgery
9. Patients on hormonal contraceptives; oral or otherwise
10. Patients on drugs, medical problems that may prolong or shorten the duration of rocuronium- (eg.. aminoglycosides, magnesium)
11. Patients with a history of allergy to rocuronium or sugammadex

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Deep block versus Moderate block: Impact on surgical satisfaction | Every 15 minutes from first laparoscopic view till the removal of laparoscopes at the end of surgery or up to 8 hours from 1st score.
  The surgeon will be required to score the quality of operating conditions every 15 minutes from 1st visualisation of peritoneal cavity until the removal of laparoscopes at the end of surgery.

SECONDARY OUTCOMES:
Deep block versus Moderate block: Patient satisfaction score | Post Anesthetic Recovery Score done at half hour from time of arrival at PACU and patient deemed fit for discharge up to 2 hours from time of arrival at PACU
  A blinded recovery nurse will administer Patient Satisfaction Questionaire
Deep block versus Moderate block: Pain score | Post Anesthetic Recovery Score done at half hour from time of arrival at PACU and patient deemed fit for discharge up to 2 hours from time of arrival at PACU
  A blinded recovery nurse will obtain the Pain Score using Visual Analogue Scale
Deep block versus Moderate block: PONV Score | Post Anesthetic Recovery Score done at half hour from time of arrival at PACU and patient deemed fit for discharge up to 2 hours from time of arrival at PACU
  A blinded recovery nurse will obtain the PONV Score using 4 point PONV scoring

CONTACTS AND LOCATIONS:
Overall Officials: Vanitha Sivanaser, M.Med Anaes (UM), Principal Investigator — Kuala Lumpur General Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Song D, Joshi GP, White PF. Fast-track eligibility after ambulatory anesthesia: a comparison of desflurane, sevoflurane, and propofol. Anesth Analg. 1998 Feb;86(2):267-73. doi: 10.1097/00000539-199802000-00009. PMID 9459231
- [Background] Gupta A, Stierer T, Zuckerman R, Sakima N, Parker SD, Fleisher LA. Comparison of recovery profile after ambulatory anesthesia with propofol, isoflurane, sevoflurane and desflurane: a systematic review. Anesth Analg. 2004 Mar;98(3):632-41, table of contents. doi: 10.1213/01.ane.0000103187.70627.57. PMID 14980911
- [Background] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482
- [Background] Geldner G, Niskanen M, Laurila P, Mizikov V, Hubler M, Beck G, Rietbergen H, Nicolayenko E. A randomised controlled trial comparing sugammadex and neostigmine at different depths of neuromuscular blockade in patients undergoing laparoscopic surgery. Anaesthesia. 2012 Sep;67(9):991-8. doi: 10.1111/j.1365-2044.2012.07197.x. Epub 2012 Jun 14. PMID 22698066
- [Background] Woo T, Kim KS, Shim YH, Kim MK, Yoon SM, Lim YJ, Yang HS, Phiri P, Chon JY. Sugammadex versus neostigmine reversal of moderate rocuronium-induced neuromuscular blockade in Korean patients. Korean J Anesthesiol. 2013 Dec;65(6):501-7. doi: 10.4097/kjae.2013.65.6.501. Epub 2013 Dec 26. PMID 24427455
- [Background] Carron M, Veronese S, Foletto M, Ori C. Sugammadex allows fast-track bariatric surgery. Obes Surg. 2013 Oct;23(10):1558-63. doi: 10.1007/s11695-013-0926-y. PMID 23519634
- [Background] Jones RK, Caldwell JE, Brull SJ, Soto RG. Reversal of profound rocuronium-induced blockade with sugammadex: a randomized comparison with neostigmine. Anesthesiology. 2008 Nov;109(5):816-24. doi: 10.1097/ALN.0b013e31818a3fee. PMID 18946293
- [Background] Della Rocca G, Pompei L, Pagan DE Paganis C, Tesoro S, Mendola C, Boninsegni P, Tempia A, Manstretta S, Zamidei L, Gratarola A, Murabito P, Fuggiano L, DI Marco P. Reversal of rocuronium induced neuromuscular block with sugammadex or neostigmine: a large observational study. Acta Anaesthesiol Scand. 2013 Oct;57(9):1138-45. doi: 10.1111/aas.12155. Epub 2013 Jul 14. PMID 23849107
- [Background] Gaszynski T, Szewczyk T, Gaszynski W. Randomized comparison of sugammadex and neostigmine for reversal of rocuronium-induced muscle relaxation in morbidly obese undergoing general anaesthesia. Br J Anaesth. 2012 Feb;108(2):236-9. doi: 10.1093/bja/aer330. Epub 2011 Oct 19. PMID 22012861
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Vender JS, Gray J, Landry E, Gupta DK. Intraoperative acceleromyography monitoring reduces symptoms of muscle weakness and improves quality of recovery in the early postoperative period. Anesthesiology. 2011 Nov;115(5):946-54. doi: 10.1097/ALN.0b013e3182342840. PMID 21946094
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear T, Vender JS, Gray J, Landry E. Postoperative residual neuromuscular blockade is associated with impaired clinical recovery. Anesth Analg. 2013 Jul;117(1):133-41. doi: 10.1213/ANE.0b013e3182742e75. Epub 2013 Jan 21. PMID 23337416
- [Background] Apfel CC, Roewer N, Korttila K. How to study postoperative nausea and vomiting. Acta Anaesthesiol Scand. 2002 Sep;46(8):921-8. doi: 10.1034/j.1399-6576.2002.460801.x. PMID 12190791
- [Background] White H, Black RJ, Jones M, Mar Fan GC. Randomized comparison of two anti-emetic strategies in high-risk patients undergoing day-case gynaecological surgery. Br J Anaesth. 2007 Apr;98(4):470-6. doi: 10.1093/bja/aem001. Epub 2007 Feb 22. PMID 17317757